CLINICAL TRIAL: NCT05669456
Title: Zeit Alert for Stroke at Home (ZASH) Protocol
Acronym: ZASH
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Zeit Medical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ZM-OP2
Record Dates: First submitted 2022-12-11; First posted 2022-12-30 (Actual); Last update posted 2022-12-30 (Actual); Status verified 2022-12

CONDITIONS: Acute Ischemic Stroke; Ischemic Stroke; Stroke
Keywords: reoccurring; detection
MeSH Terms: conditions — Ischemic Stroke; Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Halo Alert System — The Halo Alert System consists of an EEG sensor headband and is paired with a data transfer device.

SUMMARY:
This is a single-arm, observational, feasibility study to evaluate if the Halo Alert System can be used in the future to detect stroke events in individuals at risk for stroke wearing the Halo Alert System overnight.

DETAILED DESCRIPTION:
This is a single-arm, observational, feasibility study to evaluate if the Halo Alert System can be used in the future to detect stroke events in individuals at risk for stroke wearing the Halo Alert System overnight. The Halo Alert System consists of an EEG sensor headband and is paired with a data transfer device. Approximately 300 subjects with elevated stroke risk will be enrolled and followed for a duration of 90 days. The EEG tracing for each study subject will be labeled after study conclusion with the help of clinically available information on the occurrence of a recurrent stroke. The labeled data will then be used to further develop the existing (operating room based) stroke detection algorithm and adjust the algorithm for outpatient use.

ELIGIBILITY:
Inclusion Criteria:

1. New ischemic stroke confirmed by neuroimaging (CT or MRI scans) as the reason for current hospital admission or stroke clinics visit. Time from ictus to enrollment should be ≤ 2 weeks;
2. RRE-90 > 2;
3. Age ≥ 18 years old;
4. Patient is discharged to home;
5. Provision of signed and dated informed consent form.

Exclusion Criteria:

1. Subject is a member of a vulnerable population, such as prisoners, individuals without legal papers, or otherwise exploitable population;
2. Treatment with another investigational drug or intervention within the last two (2) weeks prior to start of this study, if said drug/intervention is expected to interfere with the normal function of the Halo Alert System;
3. Does not have WIFI internet access in their home;
4. Does not have access to a smartphone;
5. Open traumatic injury on the head;
6. Allergy to any of the components of the headband, such as the fabric of the band (88% Rayon, 9% Nylon, 3% Spandex), the electrode surfaces (conductive silver ink.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes subjects who are 18 years of age or older with a new acute ischemic stroke confirmed by neuroimaging (CT or MRI scans) as the primary reason for hospital or clinic presentation during which screening took place.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Halo Alert System to collect EEG data for algorithm development | 12 months enrollment period
  Subject's data collection with the Halo Alert System to assess the feasibility of EEG based stroke detection at home for algorithm development.

IPD SHARING:
Plan to Share IPD: No